CLINICAL TRIAL: NCT01998139
Title: Endothelial Microparticles as a Biomarker for Diagnosis and Prognosis in Early Sepsis
Status: Completed | Type: Observational
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: Hamad Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 1305013944; NPRP 6-1348-3-321 (Other: Qatar National Research Fund); 13-00309 (Other: JIRB)
Record Dates: First submitted 2013-11-22; First posted 2013-11-28 (Estimated); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Systemic Inflammatory Response Syndrome
MeSH Terms: conditions — Systemic Inflammatory Response Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test Cohort: EMP levels will be measured at ICU admission in subjects with physician-suspected sepsis. For each subject, the final diagnosis of sepsis or non-sepsis critical illness will be adjudicated using standard criteria. The subjects without sepsis will form the Test Cohort.
- Validation Cohort: EMP levels will be measured at ICU admission in subjects with physician-suspected sepsis. For each subject, the final diagnosis of sepsis or non-sepsis critical illness will be adjudicated using standard criteria.The subjects determined to have sepsis will serve as the Validation Cohort .

SUMMARY:
Sepsis is a major global health problem, leading to substantial morbidity and mortality despite medical care. The initial diagnosis of sepsis is a clinical challenge, as it is based on nonspecific systemic criteria. Excessive endothelial activation is a cardinal feature of sepsis and contributes to microvascular leak, edema, circulatory shock and organ failure. Activated endothelial cells shed endothelial microparticles (EMPs) which can be measured in plasma and are found at low levels in healthy subjects. Elevated EMPs have been reported in sepsis, but whether their effect is beneficial or deleterious is unclear. In this context, we hypothesize that circulating EMP levels can be assessed as a biomarker differentiating sepsis from non-sepsis critical illness. This may also suggest that EMP levels correlate with 30-day mortality. We propose to measure circulating EMPs at ICU admission in subjects with suspected sepsis. Final diagnoses will be adjudicated using standard criteria and 30-day mortality ascertained. Subjects determined not to have sepsis will serve as the control group. EMP levels will be correlated with diagnosis to ascertain the utility of EMP levels as a diagnostic biomarker for sepsis. For those subjects with proven sepsis, EMP levels will be correlated to 30-day mortality to assess EMP level as a prognostic marker in sepsis.

DETAILED DESCRIPTION:
In the presence of infection, normal immune and physiologic responses act in concert to eradicate pathogens. When these responses are inappropriately regulated, sepsis develops. Sepsis is characterized by systemic manifestations of infection. The diagnosis is made by identifying at least 2 of the components of the systemic inflammatory response syndrome (SIRS), based on four clinical and laboratory criteria: respiratory rate, tachycardia, temperature, and leukocyte level in the presence of a documented infection. The presence of acute organ dysfunction in this setting defines severe sepsis, and hypotension that is not reversed with fluid administration defines the entity of septic shock. Severe sepsis as well as its most severe form, septic shock, are significant global health concerns, afflicting millions of patients worldwide, increasing in incidence, and having an associated mortality rate of >25%. In the United States alone, an estimated 750,000 people develop sepsis or severe sepsis each year, and sepsis/septic shock is the 11th leading illness leading to mortality in the US. The annual cost burden of sepsis is estimated to be more than $17 billion. For these reasons, clinical investigators interested in sepsis have directed efforts toward identifying a biomarker that would be useful in making an early diagnosis of sepsis. In addition to early diagnosis, biomarkers for prognosis have been sought to guide severity assessment and to guide more personalized treatment of individual patients.

Endothelial Activation in Sepsis Endothelial activation occurs early in systemic infections and is an adaptive response, allowing leukocyte migration to sites of microbial invasion. In sepsis, however, endothelial activation is excessive and poses the following risks: harm via tissue damage due to excessive leukocyte recruitment, disseminated intravascular coagulation (DIC) relating to loss of endothelial anticoagulant properties, apoptotic death of endothelial cells, and loss of microvascular barrier function. The dysfunctional endothelial barrier leads to vascular leak and tissue edema, hallmarks of sepsis. This loss of endothelial barrier function is linked to increased morbidity and mortality in animal models of sepsis.

Endothelial Microparticles Microparticles are intact vesicles of a size 0.2-2.0 μm which are released from plasma membranes of multiple cell types in the setting of cell injury, activation, and/or apoptosis. In healthy individuals, microparticles found in the plasma are derived from platelets, erythrocytes, leukocytes, and endothelial cells. EMPS generally circulate at a relatively low level and reflect normal endothelial cell turnover. Elevated circulating levels of EMPs can be identified in a number of illnesses including sickle cell disease, immune-mediated thrombotic syndromes such as antiphospholipid syndrome and heparin-induced thrombocytopenia, diabetes, chronic renal failure, acute coronary syndrome, stroke, venous thromboembolic disease, metabolic syndrome, severe hypertension, paroxysmal nocturnal hemoglobinuria, and multiple sclerosis. The functional roles that may be played by endothelial microparticles are diverse and include neutrophil activation, chemotactic attraction of leukocytes, platelet aggregation, generation of thrombin (in vitro) and superoxide anions, stimulation of endothelial proliferation, induction of angiogenesis, MMP-2 and MMP-9 expression enabling vascular invasion of the basement membrane, and carrying of endothelial proteins and protein C.

Given the importance of the endothelium in the pathogenesis of sepsis, we propose to examine the role of endothelial-derived microparticles (EMPs) as a biomarker in sepsis.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18 and older
* Clinician-suspected diagnosis of sepsis
* Willingness of subject or Legally Authorized Representative (LAR) to participate in the study

Exclusion Criteria:

* Desire to forego life-sustaining therapy
* Trauma or surgical subjects
* Pregnancy
* Subjects who, in the opinion of the treating physician and/or investigator, would be at increased risk by the additional blood draw, for instance, subjects with severe anemia, or subjects with anemia who are unwilling or unable to receive blood transfusions

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be eligible for enrollment at the time of clinician decision to admit to the Medical Intensive Care Unit (MICU) for presumed sepsis.
Sampling Method: Probability Sample
Enrollment: 137 (Actual)
Dates: Start 2013-07 (Actual); Primary Completion 2019-02 (Actual); Study Completion 2019-02 (Actual)

PRIMARY OUTCOMES:
EMP level as predictive biomarker for diagnosis of sepsis. | 5 days
  To evaluate the hypothesis that EMP level is a predictive biomarker for the diagnosis of sepsis. For the primary objective, a prospective, cross-sectional, case control design will be utilized. EMP levels will be measured at ICU admission in subjects with physician-suspected sepsis. For each subject, the final diagnosis of sepsis or non-sepsis critical illness will be adjudicated using standard criteria, and the subjects determined to have sepsis will serve as the cases while those subjects without sepsis will form the control group.

SECONDARY OUTCOMES:
EMP level as a predictive biomarker for mortality in sepsis. | 30 days
  To evaluate the hypothesis that EMP level is a predictive biomarker for mortality in sepsis. For the secondary objective, EMP levels will be measured on admission and daily for the first 5 ICU days or until the subject dies or leaves the ICU. While data will be collected prospectively on all subjects, the cohort for analysis for this objective will include only those subjects with a validated diagnosis of sepsis. In these subjects, 30-day mortality will be ascertained, and EMP levels correlated with mortality to determine the utility of EMPs as a biomarker for mortality risk in sepsis.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald G Crystal, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (2):
- Weill Cornell Medical College, New York, New York, United States
- Hamad Medical Corporation, Doha, Qatar

IPD SHARING:
Plan to Share IPD: Undecided